CLINICAL TRIAL: NCT02949557
Title: A Comparative Clinical and Radiographic Evaluation of Demineralized Freeze Dried Bone Allograft (DFDBA) and Xenograft (Cerabone)TM With Decortication in the Treatment of Periodontal Intraosseous Defects
Brief Title: DFDBA and Xenograft (Cerabone)TM With Decortication in Intrabony Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_54500
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-08

CONDITIONS: Periodontal Intrabony Defects
MeSH Terms: interventions — Cerebral Decortication; Bone Transplantation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decortication +DFDBA (Active Comparator): After phase 1 therapy patients were assigned for decortication+ DFDBA group. Mucoperiosteal flaps were reflected. After open flap debridement, decortication was performed and DFDBA graft was placed in the treatment of intrabony defects.
  Interventions: Procedure: Decortication + bone grafts
- Decortication+ Xenograft (Cerabone)TM (Active Comparator): After phase 1 therapy patients were assigned for decortication+ xenograft (Cerabone)TM group. Mucoperiosteal flaps were reflected. After open flap debridement, decortication was performed and DFDBA graft was placed in the treatment of intrabony defects.
  Interventions: Procedure: Decortication + bone grafts

INTERVENTIONS:
Procedure: Decortication + bone grafts

SUMMARY:
DFDBA is an allograft that possesses osteoconductive and osteoinductive properties. It has the potential for osteoinduction due to increased expression of bone morphogenetic protein (BMP).Cerabone™ has shown maximum resemblance to human bone with the potential to reconstruct bone defects. Decortication is performed as a part of guided bone regeneration (GBR) procedure as it enhances the healing process.Therefore a combination of decortication and bone graft when applied in periodontal intrabony defect would enhance the regeneration of periodontium.

DETAILED DESCRIPTION:
There have been great strides in the management of periodontal intrabony defects, especially with the use of bone graft materials. It is necessary to choose the most appropriate material and procedure in order to obtain the desired regeneration. Among the bone grafts, Demineralised freezed dried bone allograft (DFDBA) and xenografts have shown good results in the management of intrabony defects. Recently, a novel bovine xenograft i.e., Cerabone™ has shown maximum resemblance to human bone with the potential to reconstruct bone defects. Decortication or intramarrow penetration of the bone has shown favourable results in guided bone regeneration procedures. So the goal of the present study was to check the efficacy of decortication with decalcified freeze dried bone allograft (DFDBA) and Cerabone™ bone grafts and to compare the response between the bonegrafts placed following decortication using RVG and CBCT, in intrabony defect.

The combination of decortication with bone grafts i.e., DFDBA and (Cerabone)TM can be an added advantage in the treatment of intrabony defects. To the best of the investigators knowledge no clinical trial reports this combination therapy in scientific literature. There is need for further research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Age group 25-45 years
* Moderate periodontitis with pocket probing depth more than 5 mm
* Bilaterally similiar intrabony defects
* systemically healthy patients
* Good compliance

Exclusion Criteria:

* medically compromised
* Pregnant and lactating women
* Smoking
* teeth with mobility and furcation involvement

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
clinical attachment level | 9 months
  clinical attachment level measured in mm from cementoenamel junction to the base of the pocket
Bone fill | 9 months
  Bone fill measured in mm in radiographs from alveolar crest to base of the pocket
Pocket probing depth | 9 months
  pocket probing depth level measured in mm from gingival margin to base of the pocket

SECONDARY OUTCOMES:
Plaque Index (PI) | 9 month
  Plaque index is measured for periodontal health
Periodontal disease index | 9 months
  Periodontal disease index is measured for periodontal health
Gingival Bleeding Index | 9 months
  Gingival bleeding index is measured for periodontal health